CLINICAL TRIAL: NCT03052322
Title: A Multicenter, Randomized, Double-blind, Phase III Trial to Evaluate the Safety, Immunogenicity, and Efficacy of MSB11022 Compared With Humira® in Patients With Moderately to Severely Active Rheumatoid Arthritis
Brief Title: MSB11022 in Moderate to Severe Rheumatoid Arthritis
Acronym: Auriel-RA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fresenius Kabi SwissBioSim GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS200588-0004; 2016-002852-26 (EudraCT Number)
Record Dates: First submitted 2017-01-29; First posted 2017-02-14 (Actual); Results first posted 2019-04-23 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Moderate to Severe Rheumatoid Arthritis
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MSB11022 (Experimental)
  Interventions: Drug: MSB11022
- EU-Humira (Active Comparator)
  Interventions: Drug: EU-Humira

INTERVENTIONS:
Drug: MSB11022 — Participants received MSB11022 (modified buffer and stabilizer) subcutaneously at dose of 40 milligram (mg) every other week from Day 1 up to Week 48.
  Other Names: Adalimumab
  Arms: MSB11022
Drug: EU-Humira — Participants received EU-Humira subcutaneously at dose of 40 mg every other week from Day 1 up to Week 48.
  Arms: EU-Humira

SUMMARY:
The purpose of this study is to compare the efficacy, safety and immunogenicity of MSB11022 and Humira® in adult participants with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis based on 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) criteria
* At least 6 tender (of 68 assessed) and 6 swollen (of 66 assessed) joints at screening and baseline
* Must have received methotrexate for at least 12 weeks and been on a stable dose for at least 4 weeks prior to the first study dose
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Evidence of untreated or inadequately treated latent or active Tuberculosis
* Evidence of uncontrolled, clinically significant diseases
* Any second disease-modifying antirheumatic drugs must be washed out prior to the first study dose
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Fresenius Kabi SwissBioSim GmbH
Locations (46):
- Bulgaria (12):
  - MHAT "Trimontium", OOD, Plovdiv
  - MHAT-Plovdiv AD, Plovdiv
  - UMHAT "Kaspela", EOOD, Plovdiv
  - Medical Center "Teodora", EOOD, Rousse
  - MHAT - Ruse, AD, Rousse
  - MHAT - Shumen, AD, Shumen
  - MHAT "Lyulin", EAD, Sofia
  - Medical Center "Excelsior", OOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - DCC 17 - Sofia EOOD, Sofia
  - Military Medical Academy - MHAT - Sofia, Sofia
  - MC "Synexus - Sofia", EOOD, Sofia
- Czechia (10):
  - Revmatologie Bruntal, s.r.o., Bruntál
  - Ccbr-Synarc A/S, Ostrava
  - A-SHINE s.r.o., Pilsen
  - CLINTRIAL s.r.o., Prague
  - Revmatologicky Ustav, Prague
  - Nuselska poliklinika, Prague
  - Revma Praha, s.r.o., Prague
  - Revmatologicka ambulance, Praha 4 Nusle
  - MEDICAL PLUS s.r.o., Uherské Hradiště
  - PV - Medical, s.r.o., Zlín
- Germany (2):
  - Studienambulanz Dr. Wassenberg, Ratingen, North Rhine-Westphalia
  - HRF Hamburger Rheuma Forschungszentrum, Hamburg
- Hungary (7):
  - Dr. Kenessey Albert Korhaz-Rendelointezet, Balassagyarmat
  - Revita Reumatologiai Rendelo, Budapest
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - DRC Szekesfehervar, Székesfehérvár
  - Mentahaz Maganorvosi Kozpont, Székesfehérvár
  - Vital Medical Center, Veszprém
  - Synexus Magyarorszag Egeszsegugyi Szolgaltato Kft.- Zalaegerszeg AS, Zalaegerszeg
- Poland (13):
  - KLIMED Marek Klimkiewicz, Bialystok
  - ClinicMed Badurski i wspolnicy Spolka Jawna, Bialystok
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Centrum Medyczne Angelius Provita, Katowice
  - Malopolskie Centrum Medyczne s.c., Krakow
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska sp. komandytowo-akcyjna, Lodz
  - RCMed, Nowy Duninów
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
  - Niepubliczny Zaklad Opieki Zdrowotnej "Nasz Lekarz" Praktyka Grupowa Lekarzy Rodzinnych z, Torun
  - Medycyna Kliniczna, Warsaw
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - Niepubliczny Zakład Opieki Zdrowotnej "Biogenes" Sp. z o.o., Wroclaw
  - KLIMED Marek Klimkiewicz, Łomża
- United Kingdom (2):
  - Glasgow Royal Infirmary, Glasgow, Strathclyde
  - Whipps Cross University Hospital, London

REFERENCES:
- [Derived] Huizinga TWJ, Torii Y, Muniz R. Adalimumab Biosimilars in the Treatment of Rheumatoid Arthritis: A Systematic Review of the Evidence for Biosimilarity. Rheumatol Ther. 2021 Mar;8(1):41-61. doi: 10.1007/s40744-020-00259-8. Epub 2020 Dec 1. PMID 33263165

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in 1:1 ratio to receive either MSB11022 or EU-Humira for 48 weeks.
Period: Overall Study
Arm/Group | MSB11022 | EU-Humira
Started | 143 | 145
Completed | 122 | 113
Not Completed | 21 | 32
Not completed — Other un-specified | 1 | 2
Not completed — Withdrawal by Subject | 10 | 9
Not completed — Death | 0 | 2
Not completed — Lack of Efficacy | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 2 | 4
Not completed — Adverse Event | 6 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MSB11022 | EU-Humira | Total
Number analyzed (Participants) | 143 | 145 | 288
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.9 (11.9) | 54.0 (11.0) | 53.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 119 | 227
  Male | 35 | 26 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 140 | 144 | 284
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 142 | 143 | 285
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events of Special Interest (AESI)
Description: Adverse event (AE) was defined as any untoward medical occurrence in participants, which does not necessarily have causal relationship with treatment. Term Treatment-emergent Adverse Events (TEAE) is defined as AEs starting/worsening after first intake of the study drug. Hypersensitivity was the pre-defined TEAE of special Interest for this study. The percentage of participants with treatment emergent AESIs (hypersensitivity) were reported.
Time Frame: Up to Week 52
Population: The Safety Analysis Set included all randomized participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Percentage of Participants | 4.2 [1.6 to 8.9] | 5.5 [2.4 to 10.6]

2. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 20 (ACR20) Response at Week 12
Description: The ACR 20 Response is defined as greater than or equal to (>=) 20 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=20 percent improvement in 3 of following 5 assessments: participant's assessment of pain using Visual Analog Scale (VAS ; 0-10 millimeter [mm], 0 mm=no pain and 10 mm=worst possible pain), participant's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas). The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and acute-phase marker (CRP).
Time Frame: Week 12
Population: Intent-To-Treat (ITT) Analysis Set included all participants randomly allocated to a treatment, based on intent to treat "as randomized" principle (planned treatment regimen rather than actual treatment given in case of any difference). Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 142 | 141
Percentage of Participants | 79.6 [72.0 to 85.9] | 80.9 [73.4 to 86.9]

3. Secondary Outcome: Percentage of Participants With Positive Anti-Drug Antibodies (ADAs) Status to Adalimumab
Description: Percentage of participants with positive anti-Drug antibodies (ADAs) status to Adalimumab were reported.
Time Frame: Baseline, Week 2, 4, 12, 24, 36 and 52
Population: The Safety Analysis Set included all randomized participants who received at least one dose of study treatment. Here "Number analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Number; unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Percentage of Participants
  Baseline: number analyzed (Participants) | 142 | 144
  Baseline | 7.7 | 4.2
  Week 2 | 20.3 | 15.2
  Week 4: number analyzed (Participants) | 141 | 141
  Week 4 | 29.8 | 21.3
  Week 12: number analyzed (Participants) | 142 | 140
  Week 12 | 54.2 | 48.6
  Week 24: number analyzed (Participants) | 139 | 133
  Week 24 | 71.9 | 61.7
  Week 36: number analyzed (Participants) | 124 | 121
  Week 36 | 66.9 | 65.3
  Week 52: number analyzed (Participants) | 120 | 119
  Week 52 | 60.8 | 62.2

4. Secondary Outcome: Anti-Drug Antibodies (ADAs) Titer Levels for Adalimumab
Description: Titer was defined as the degree to which the antibody-serum sample could be diluted and still contained detectable amounts of antibody. Anti-Drug Antibodies (ADAs) titers for adalimumab was reported. Data was collected using validated bioanalytical method.
Time Frame: Baseline, Week 2, 4, 12, 24, 36 and 52
Population: The Safety Analysis Set included all randomized participants who received at least one dose of study treatment. Here "Number of participants analyzed" signifies those who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at specified time points.
Measure: Median (Full Range); unit: Titer
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 115 | 104
Titer
  Baseline: number analyzed (Participants) | 11 | 6
  Baseline | 4.0 [1 to 512] | 1.5 [1 to 8]
  Week 2: number analyzed (Participants) | 29 | 22
  Week 2 | 4.0 [1 to 32768] | 12.0 [1 to 1024]
  Week 4: number analyzed (Participants) | 42 | 30
  Week 4 | 6.0 [1 to 16384] | 6.0 [1 to 512]
  Week 12: number analyzed (Participants) | 77 | 68
  Week 12 | 16.0 [1 to 4096] | 16.0 [1 to 16384]
  Week 24: number analyzed (Participants) | 100 | 82
  Week 24 | 16.0 [1 to 32768] | 24.0 [1 to 131072]
  Week 36: number analyzed (Participants) | 83 | 79
  Week 36 | 16.0 [1 to 32768] | 16.0 [1 to 131072]
  Week 52: number analyzed (Participants) | 73 | 74
  Week 52 | 16.0 [1 to 16384] | 12.0 [1 to 32768]

5. Secondary Outcome: Percentage of Participants With Confirmed Neutralizing Antibodies (NAb) Status to Adalimumab
Description: Percentage of participants with confirmed neutralizing antibodies status to Adalimumab were reported.
Time Frame: Baseline, Week 2, 4, 12, 24, 36 and 52
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 115 | 104
Percentage of Participants
  Baseline: number analyzed (Participants) | 11 | 6
  Baseline | 45.5 | 50.0
  Week 2: number analyzed (Participants) | 29 | 22
  Week 2 | 31.0 | 40.9
  Week 4: number analyzed (Participants) | 42 | 30
  Week 4 | 33.3 | 30.0
  Week 12: number analyzed (Participants) | 77 | 68
  Week 12 | 33.8 | 38.2
  Week 24: number analyzed (Participants) | 100 | 82
  Week 24 | 27.0 | 29.3
  Week 36: number analyzed (Participants) | 83 | 79
  Week 36 | 24.1 | 29.1
  Week 52: number analyzed (Participants) | 73 | 74
  Week 52 | 32.9 | 39.2

6. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 20 (ACR20) Response at Week 2, 4, 8, 24 and 52
Description: The ACR 20 Response is defined as greater than or equal to (>=) 20 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=20 percent improvement in 3 of following 5 assessments: patient's assessment of pain using Visual Analog Scale (VAS ; 0-10 millimeter [mm], 0 mm=no pain and 10 mm=worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas). The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and acute-phase marker (CRP).
Time Frame: Week 2, 4, 8, 24 and 52
Population: ITT Analysis Set included all participants randomly allocated to a treatment, based on intent to treat "as randomized" principle (planned treatment regimen rather than actual treatment given in case of any difference). Here "Number analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Percentage of Participants
  Week 2 | 30.0 [22.55 to 38.32] | 29.7 [22.36 to 37.80]
  Week 4: number analyzed (Participants) | 142 | 144
  Week 4 | 52.1 [43.58 to 60.56] | 52.8 [44.29 to 61.15]
  Week 8: number analyzed (Participants) | 142 | 144
  Week 8 | 71.1 [62.93 to 78.42] | 72.9 [64.89 to 79.98]
  Week 24: number analyzed (Participants) | 139 | 133
  Week 24 | 88.5 [81.98 to 93.28] | 83.3 [75.86 to 89.25]
  Week 52: number analyzed (Participants) | 122 | 119
  Week 52 | 81.8 [73.78 to 88.24] | 86.4 [78.92 to 92.05]

7. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 50 (ACR50) Response at Week 2, 4, 8, 12, 24 and 52
Description: The ACR 50 Response is defined as greater than or equal to (>=) 50 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=50 percent improvement in 3 of following 5 assessments: patient's assessment of pain using Visual Analog Scale (VAS ; 0-10 millimeter [mm], 0 mm=no pain and 10 mm=worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas). The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and acute-phase marker (CRP).
Time Frame: Week 2, 4, 8, 12, 24 and 52
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Percentage of Participants
  Week 2 | 6.4 [2.9 to 11.9] | 6.2 [2.9 to 11.5]
  Week 4: number analyzed (Participants) | 142 | 144
  Week 4 | 17.6 [11.7 to 24.9] | 19.4 [13.3 to 26.9]
  Week 8: number analyzed (Participants) | 142 | 144
  Week 8 | 40.8 [32.7 to 49.4] | 34.7 [26.9 to 43.1]
  Week 12: number analyzed (Participants) | 142 | 141
  Week 12 | 54.2 [45.7 to 62.6] | 51.1 [42.5 to 59.6]
  Week 24: number analyzed (Participants) | 139 | 133
  Week 24 | 65.5 [56.9 to 73.3] | 60.6 [51.7 to 68.9]
  Week 52: number analyzed (Participants) | 122 | 119
  Week 52 | 64.5 [55.3 to 72.9] | 66.1 [56.8 to 74.6]

8. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 70 (ACR70) Response at Week 2, 4, 8, 12, 24 and 52
Description: The ACR 70 Response is defined as greater than or equal to (>=) 70 percent improvement in swollen joint count (66 joints) and tender joint count (68 joints) and >=70 percent improvement in 3 of following 5 assessments: patient's assessment of pain using Visual Analog Scale (VAS ; 0-10 millimeter [mm], 0 mm=no pain and 10 mm=worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain]), physician's global assessment of disease activity using VAS, participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas). The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and acute-phase marker (CRP).
Time Frame: Week 2, 4, 8, 12, 24 and 52
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Percentage of Participants
  Week 2 | 0.7 [0.0 to 3.9] | 0.7 [0.0 to 3.8]
  Week 4: number analyzed (Participants) | 142 | 144
  Week 4 | 4.9 [2.0 to 9.9] | 2.8 [0.8 to 6.9]
  Week 8: number analyzed (Participants) | 142 | 144
  Week 8 | 14.8 [9.4 to 21.7] | 12.5 [7.6 to 19.0]
  Week 12: number analyzed (Participants) | 142 | 141
  Week 12 | 26.8 [19.7 to 34.8] | 19.9 [13.6 to 27.4]
  Week 24: number analyzed (Participants) | 139 | 133
  Week 24 | 33.8 [26.0 to 42.3] | 35.6 [27.5 to 44.4]
  Week 52: number analyzed (Participants) | 122 | 119
  Week 52 | 39.7 [30.9 to 48.9] | 42.4 [33.3 to 51.8]

9. Secondary Outcome: Change From Baseline in Disease Activity Score Based on a 28 Joint Count- Erythrocyte Sedimentation Rate (DAS28-ESR) Score at Week 2, 4, 8, 12, 24 and 52
Description: DAS calculated on 28 joints is composite score derived from 4 measures: number of swollen joints (out of 28), number of tender joints (out of 28), Erythrocyte sedimentation rate (ESR), Patient's Global Assessment of Disease Activity on visual analog scale (VAS). Overall disease activity score DAS28 was derived using following formulas from DAS28:DAS28=0.56*√(TJC28)+0.28*√(SJC28) + 0.014*GH+0.70*ln(ESR). Where: TJC28 = 28 joint count for tenderness, SJC28 = 28 joint count for swelling, ln(ESR) = natural log of ESR, GH = general health component of DAS (ie, Patient's Global Assessment of Disease Activity, assessed using scale of 1-100 where 100 is maximal activity); For analyses, GH divided by 10 & converted to 0.5 scale, i.e, 0, 0.5, 1, 1.5. DAS28-ESR of >5.1 implies active disease, <3.2 low disease activity, & <2.6 remission. Change of 1.2(twice measurement error)=significant change of disease activity state. Overall score ranges from 0-10 where higher score means more severe disease.
Time Frame: Baseline, Week 2, 4, 8, 12, 24 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Units on a scale
  Change at Week 2: number analyzed (Participants) | 140 | 145
  Change at Week 2 | -0.9 (0.9) | -0.7 (0.9)
  Change at Week 4: number analyzed (Participants) | 141 | 144
  Change at Week 4 | -1.4 (1.1) | -1.2 (1.0)
  Change at Week 8: number analyzed (Participants) | 142 | 144
  Change at Week 8 | -1.9 (0.9) | -1.7 (1.1)
  Change at Week 12: number analyzed (Participants) | 142 | 141
  Change at Week 12 | -2.4 (1.1) | -2.1 (1.2)
  Change at Week 24: number analyzed (Participants) | 138 | 132
  Change at Week 24 | -2.7 (1.0) | -2.3 (1.2)
  Change at Week 52: number analyzed (Participants) | 121 | 118
  Change at Week 52 | -2.8 (1.1) | -2.5 (1.1)

10. Secondary Outcome: Percentage of Participants With Disease Activity Score Based on 28-joints Count- Erythrocyte Sedimentation Rate (DAS28-ESR) Low Disease Activity and Remission at Week 2, 4, 8, 12, 24, and 52
Description: Disease Activity Score calculated on 28 joints is composite score derived from 4 measures: number of swollen joints (out of 28), -number of tender joints (out of 28), -Erythrocyte sedimentation rate (ESR), -Patient's Global Assessment of Disease Activity on visual analog scale (VAS). Overall disease activity score DAS28 was derived using following formulas from DAS28: DAS28=0.56*√(TJC28)+0.28*√(SJC28) + 0.014*GH+0.70*ln(ESR). Where: -TJC28 = 28 joint count for tenderness, -SJC28 = 28 joint count for swelling, -ln(ESR) = natural logarithm of ESR, -GH = general health component of DAS (ie, Patient's Global Assessment of Disease Activity, assessed using scale of 1 to 100 where 100 is maximal activity); For analyses, GH was divided by 10 and converted to a 0.5 scale, i.e., 0, 0.5, 1, 1.5. DAS28-ESR of >5.1 implies active disease, <3.2 low disease activity, and <2.6 remission.
Time Frame: Week 2, 4, 8, 12, 24, and 52
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Percentage of Participants
  Low Disease Activity: Week 2 | 10.0 [5.6 to 16.2] | 8.3 [4.4 to 14.0]
  Low Disease Activity: Week 4: number analyzed (Participants) | 142 | 144
  Low Disease Activity: Week 4 | 20.6 [14.2 to 28.2] | 16.0 [10.4 to 23.0]
  Low Disease Activity: Week 8: number analyzed (Participants) | 142 | 144
  Low Disease Activity: Week 8 | 33.1 [25.4 to 41.5] | 33.3 [25.7 to 41.7]
  Low Disease Activity: Week 12: number analyzed (Participants) | 142 | 141
  Low Disease Activity: Week 12 | 46.5 [38.1 to 55.0] | 42.6 [34.3 to 51.2]
  Low Disease Activity: Week 24: number analyzed (Participants) | 139 | 133
  Low Disease Activity: Week 24 | 55.1 [46.4 to 63.5] | 53.8 [44.9 to 62.5]
  Low Disease Activity: Week 52: number analyzed (Participants) | 122 | 119
  Low Disease Activity: Week 52 | 57.0 [47.7 to 65.9] | 56.8 [47.3 to 65.9]
  Remission: Week 2 | 3.6 [1.2 to 8.1] | 2.1 [0.4 to 5.9]
  Remission: Week 4: number analyzed (Participants) | 142 | 144
  Remission: Week 4 | 7.8 [3.9 to 13.5] | 6.9 [3.4 to 12.4]
  Remission: Week 8: number analyzed (Participants) | 142 | 144
  Remission: Week 8 | 18.3 [12.3 to 25.7] | 16.0 [10.4 to 23.0]
  Remission: Week 12: number analyzed (Participants) | 142 | 141
  Remission: Week 12 | 29.6 [22.2 to 37.8] | 24.1 [17.3 to 32.0]
  Remission: Week 24: number analyzed (Participants) | 139 | 133
  Remission: Week 24 | 31.2 [23.6 to 39.6] | 34.1 [26.0 to 42.8]
  Remission: Week 52: number analyzed (Participants) | 122 | 119
  Remission: Week 52 | 40.5 [31.7 to 49.8] | 36.4 [27.8 to 45.8]

11. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) Total Score at Week 2, 4, 8, 12, 24, and 52
Description: SDAI is numerical sum of 5 outcome parameters: tender & swollen joint count (based on 28-joint assessment), Patient's & Physician's Global Assessment of Disease Activity (VAS) & level of C-reactive protein (CRP)(milligram per deciliter (mg/dL), normal<1 mg/dL). SDAI was calculated based on following formula: SDAI = 28 joint count for swelling (SJC28) + 28 joint count for tenderness (TJC28)+GH+PGA+CRP Where: -GH =general health component of DAS (i.e. Patient's Global Assessment of Disease Activity, assessed using scale of 1 to 100 where 100 is maximal activity; For analyses, GH was divided by 10 & converted to 0.5 scale (0, 0.5, 1, 1.5).-PGA = Physician's Global Assessment of Disease Activity assessed using scale of 1 to 100 where 100 is maximal activity. For analyses, PGA will be divided by 10 & converted to 0.5 scale (0, 0.5, 1, 1.5). where [0-0.25] = 0, [0.25-0.75] = 0.5, [0.76-1.25] = 1, etc. The total score range is 0-86 & lower score indicates less disease activity.
Time Frame: Baseline, Week 2, 4, 8, 12, 24, and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Units on a scale
  Change at Week 2: number analyzed (Participants) | 139 | 145
  Change at Week 2 | -11.5 (10.6) | -9.1 (10.0)
  Change at Week 4: number analyzed (Participants) | 140 | 140
  Change at Week 4 | -18.0 (11.3) | -16.0 (10.9)
  Change at Week 8: number analyzed (Participants) | 141 | 144
  Change at Week 8 | -24.0 (10.6) | -21.4 (11.0)
  Change at Week 12: number analyzed (Participants) | 140 | 141
  Change at Week 12 | -27.9 (10.8) | -24.7 (10.9)
  Change at Week 24: number analyzed (Participants) | 136 | 131
  Change at Week 24 | -31.4 (11.2) | -27.8 (10.6)
  Change at Week 52: number analyzed (Participants) | 118 | 118
  Change at Week 52 | -31.5 (11.6) | -29.1 (10.8)

12. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Total Score at Week 2, 4, 8, 12, 24 and 52
Description: Clinical Disease Activity Index (CDAI) is a composite index (without acute-phase reactant) for assessing disease activity. The CDAI was calculated based on following formula: CDAI = 28 joint count for swelling (SJC28) + 28 joint count for tenderness (TJC28) + GH + PGA. Where, -GH = general health component of the DAS (i.e., Patient's Global Assessment of Disease Activity, assessed using a scale of 1 to 100 where 100 is maximal activity; for analyses, GH was divided by 10 and converted to a 0.5 scale, i.e., 0, 0.5, 1, 1.5 etc. where [0-0.25] = 0, [0.25-0.75] = 0.5, [0.76-1.25] = 1, etc.). -PGA = Physician's Global Assessment of Disease Activity assessed using a scale of 1 to 100 where 100 is maximal activity. For analyses, PGA was divided by 10 and converted to a 0.5 scale, ie, 0, 0.5, 1, 1.5 etc. where [0-0.25] = 0, [0.25-0.75] = 0.5, [0.76-1.25] = 1, etc. The CDAI ranges from 0 to 76. Lower score indicates less disease activity.
Time Frame: Baseline, Week 2, 4, 8, 12, 24 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Units on a scale
  Change at Week 2: number analyzed (Participants) | 139 | 145
  Change at Week 2 | -10.8 (10.3) | -8.5 (9.9)
  Change at Week 4: number analyzed (Participants) | 141 | 144
  Change at Week 4 | -17.4 (11.2) | -15.2 (10.7)
  Change at Week 8: number analyzed (Participants) | 141 | 144
  Change at Week 8 | -23.5 (10.6) | -20.6 (10.9)
  Change at Week 12: number analyzed (Participants) | 141 | 141
  Change at Week 12 | -27.4 (10.5) | -24.1 (10.7)
  Change at Week 24: number analyzed (Participants) | 138 | 132
  Change at Week 24 | -30.8 (10.9) | -27.1 (10.7)
  Change at Week 52: number analyzed (Participants) | 120 | 118
  Change at Week 52 | -31.1 (11.2) | -28.5 (10.6)

13. Secondary Outcome: Percentage of Participants With American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Boolean Remission at Week 2, 4, 8, 12, 24 and 52
Description: According to Boolean-based definition of remission of ACR/EULAR, a participant must satisfy all of the following: tender joint count <= 1, swollen joint count <= 1, CRP <= 1 mg/dL, and Patient's Global Assessment of Disease Activity <= 1 (0 to 10 VAS). PGA was assessed on a 10 mm VAS ranging from 0 (very well) to 10 (very poor), where higher scores indicate worse health condition.
Time Frame: Week 2, 4, 8, 12, 24 and 52
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Percentage of Participants
  Week 2 | 0.7 [0.0 to 3.9] | 0.0 [0.0 to 2.5]
  Week 4: number analyzed (Participants) | 142 | 144
  Week 4 | 0.7 [0.0 to 3.9] | 1.4 [0.2 to 5.1]
  Week 8: number analyzed (Participants) | 142 | 144
  Week 8 | 3.5 [1.2 to 8.0] | 4.2 [1.5 to 8.9]
  Week 12: number analyzed (Participants) | 142 | 141
  Week 12 | 5.7 [2.5 to 10.9] | 12.1 [7.2 to 18.6]
  Week 24: number analyzed (Participants) | 139 | 133
  Week 24 | 11.7 [6.8 to 18.3] | 8.4 [4.3 to 14.5]
  Week 52: number analyzed (Participants) | 122 | 119
  Week 52 | 21.0 [14.1 to 29.4] | 13.6 [7.9 to 21.1]

14. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs and TEAEs Leading to Death
Description: Adverse event(AE) was defined as any untoward medical occurrence in participants which does not necessarily have causal relationship with treatment. A serious adverse event(SAE) was AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Term TEAE is defined as AEs starting/worsening after first intake of the study drug. All abnormal physical examinations occurring during the study have been reported as Adverse events. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Week 69
Population: The Safety Analysis Set included all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Percentage of Participants
  TEAEs | 58.0 | 64.1
  Serious TEAEs | 4.9 | 9.7
  TEAEs Leading to Death | 0 | 0.7

15. Secondary Outcome: Percentage of Participants With Clinically Meaningful Differences in Vital Signs
Description: Vital signs including body temperature, respiratory rate, and heart rate (after 5-minute rest) were measured. Percentage of participants with clinically meaningful abnormalities in vital signs were reported. Clinical meaningful was determined by the investigator.
Time Frame: Up to Week 52
Population: The Safety Analysis Set included all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Percentage of Participants | 0 | 0

16. Secondary Outcome: Percentage of Participants With Clinically Meaningful Differences in Laboratory Values
Description: Laboratory parameters including hematology, urinalysis, and biochemistry analysis were analyzed.
Time Frame: Up to Week 52
Population: The Safety Analysis Set included all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Percentage of Participants | 0 | 0

17. Secondary Outcome: Percentage of Participants With Clinically Significant Abnormal Values for 12-lead Electrocardiogram (ECG) at Week 12, 24, and 52
Description: Percentage of participants with clinically significant abnormal values for 12-lead electrocardiogram (ECG) at week 12, 24, and 52 were reported.
Time Frame: Week 12, 24, and 52
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Percentage of Participants
  Week 12: number analyzed (Participants) | 142 | 141
  Week 12 | 0 | 0
  Week 24: number analyzed (Participants) | 139 | 133
  Week 24 | 0 | 1.5
  Week 52: number analyzed (Participants) | 122 | 119
  Week 52 | 0 | 0.8

18. Secondary Outcome: Percentage of Participants With Anti-Nuclear Antibody (ANA) and Anti Double-stranded Deoxyribonucleic Acid (Anti-dsDNA) at Baseline, Week 24 and 52
Description: For ANA, positivity is defined as any participant with ANA titer greater than (>) 1:160 and negativity is defined as ANA titer less than (<) 1:160. For anti-ds DNA, positivity is defined as any participant with adsDNA > 15 units per milliliter (U/mL), intermediate category is defined as value between 10 U/mL to 15 U/mL and negativity is defined as adsDNA < 10 U/mL. Percentage of participants with anti-nuclear antibody (ANA) and anti double-stranded deoxyribonucleic acid (Anti-dsDNA) at baseline, week 24 and 52 were reported.
Time Frame: Baseline, Week 24 and 52
Population: The Safety Analysis Set included all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Percentage of Participants
  Baseline: ANA: Negative | 97.2 | 95.1
  Baseline: ANA: Positive | 2.8 | 4.9
  Week 24: ANA: Negative: number analyzed (Participants) | 138 | 131
  Week 24: ANA: Negative | 92.0 | 91.6
  Week 24: ANA: Positive: number analyzed (Participants) | 138 | 131
  Week 24: ANA: Positive | 8.0 | 8.4
  Week 52: ANA: Negative: number analyzed (Participants) | 118 | 111
  Week 52: ANA: Negative | 78.8 | 84.7
  Week 52: ANA: Positive: number analyzed (Participants) | 118 | 111
  Week 52: ANA: Positive | 21.2 | 15.3
  Baseline: Anti-dsDNA: Negative: number analyzed (Participants) | 141 | 141
  Baseline: Anti-dsDNA: Negative | 97.9 | 98.6
  Baseline: Anti-dsDNA: Intermediate: number analyzed (Participants) | 141 | 141
  Baseline: Anti-dsDNA: Intermediate | 1.4 | 0.7
  Baseline: Anti-dsDNA: Positive: number analyzed (Participants) | 141 | 141
  Baseline: Anti-dsDNA: Positive | 0.7 | 0.7
  Week 24: Anti-dsDNA: Negative: number analyzed (Participants) | 138 | 132
  Week 24: Anti-dsDNA: Negative | 95.7 | 96.2
  Week 24: Anti-dsDNA: Intermediate: number analyzed (Participants) | 138 | 132
  Week 24: Anti-dsDNA: Intermediate | 2.2 | 3.0
  Week 24: Anti-dsDNA: Positive: number analyzed (Participants) | 138 | 132
  Week 24: Anti-dsDNA: Positive | 2.2 | 0.8
  Week 52: Anti-dsDNA: Negative: number analyzed (Participants) | 121 | 118
  Week 52: Anti-dsDNA: Negative | 95.0 | 97.5
  Week 52: Anti-dsDNA: Intermediate: number analyzed (Participants) | 121 | 118
  Week 52: Anti-dsDNA: Intermediate | 0.8 | 1.7
  Week 52: Anti-dsDNA: Positive: number analyzed (Participants) | 121 | 118
  Week 52: Anti-dsDNA: Positive | 4.1 | 0.8

19. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) Total Score at Baseline, Weeks 12, 24 and 52
Description: The HAQ-DI is a participant-reported questionnaire that is commonly used in RA to measure disease associated disability (assessment of physical function). It consists of several questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. HAQ-DI scores range from 0 to 3. The disability section of the questionnaire scores the participant's self-perception on the degree of difficulty (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do).
Time Frame: Baseline, Weeks 12, 24 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Units on a scale
  Baseline | 1.6 (0.6) | 1.6 (0.6)
  Week 12: number analyzed (Participants) | 142 | 141
  Week 12 | 1.1 (0.6) | 1.1 (0.6)
  Week 24: number analyzed (Participants) | 139 | 132
  Week 24 | 1.0 (0.6) | 1.0 (0.6)
  Week 52: number analyzed (Participants) | 121 | 118
  Week 52 | 0.9 (0.7) | 0.9 (0.6)

20. Secondary Outcome: Short-Form Health Survey- 36 Items (SF-36) at Baseline, Week 12, 24 and 52
Description: The Short Form Health Survey (SF-36) is a validated 36-item, patient-reported indication of overall health status not specific to any age, disease or Treatment group. The SF-36 questionnaire contains 36 questions pertaining to eight subscales of health status. These eight subscales were summarized as relating to either physical health or mental health. Physical component summary (PCS) is based primarily on physical functioning, role-physical, bodily pain, and general health scales and mental component summary (MCS) encompasses vitality, social functioning, role-emotional, and mental health scales. Score from mental health, role emotional, social functioning, and vitality domains were averaged to calculate MCS. Total score range for MCS was 0-100 (100=highest level of mental functioning). Score from physical function, role physical, bodily pain, and general health domains were averaged to calculate PCS. Total score range for PCS was 0-100 (100=highest level of physical functioning).
Time Frame: Baseline, Week 12, 24 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Units on a scale
  PCS: Baseline: number analyzed (Participants) | 134 | 134
  PCS: Baseline | 30.3 (7.6) | 30.6 (7.8)
  PCS: Week 12: number analyzed (Participants) | 142 | 141
  PCS: Week 12 | 39.0 (7.9) | 38.6 (8.6)
  PCS: Week 24: number analyzed (Participants) | 139 | 132
  PCS: Week 24 | 40.5 (8.8) | 40.8 (9.1)
  PCS: Week 52: number analyzed (Participants) | 121 | 118
  PCS: Week 52 | 41.8 (9.5) | 41.6 (9.3)
  MCS: Baseline: number analyzed (Participants) | 134 | 134
  MCS: Baseline | 40.9 (13.2) | 43.4 (11.7)
  MCS: Week 12: number analyzed (Participants) | 142 | 141
  MCS: Week 12 | 47.4 (11.3) | 48.2 (11.3)
  MCS: Week 24: number analyzed (Participants) | 139 | 132
  MCS: Week 24 | 49.8 (10.8) | 48.8 (10.9)
  MCS: Week 52: number analyzed (Participants) | 121 | 118
  MCS: Week 52 | 48.0 (10.4) | 49.3 (11.5)

21. Secondary Outcome: Euro-Quality of Life - 5 Dimension-5 Levels (EQ-5D-5L) Utility Index Score at Baseline, Week 12, 24 and 52
Description: EQ-5D-5L is a standardized, participant-rated questionnaire to assess health-related quality of life. The EQ-5D-5L includes 2 components: the EQ-5D-5L health state profile (descriptive system) and the EQ-5D-5L Visual Analog Scale. The EQ-5D-5L descriptive system provides a profile of the participant's health state 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response options (no problems, slight problems, moderate problems, severe problems and extreme problems) that reflect increasing levels of difficulty. The participant was asked to indicate his/her current health state by selecting the most appropriate level in each of the 5 dimensions. Responses to the 5 dimension scores were combined and converted into a single preference-weighted health utility index score 0 (0.0- worst health state) to 1 (1.0- better health state) representing the general health status of the individual based on the UK scoring algorithm.
Time Frame: Baseline, Week 12, 24 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Units on a scale
  Baseline: number analyzed (Participants) | 134 | 133
  Baseline | 0.6 (0.2) | 0.6 (0.2)
  Week 12: number analyzed (Participants) | 142 | 140
  Week 12 | 0.8 (0.1) | 0.8 (0.1)
  Week 24: number analyzed (Participants) | 139 | 132
  Week 24 | 0.8 (0.1) | 0.8 (0.1)
  Week 52: number analyzed (Participants) | 121 | 118
  Week 52 | 0.8 (0.2) | 0.8 (0.1)

22. Secondary Outcome: Euro-Quality of Life - 5 Dimension-5 Levels (EQ-5D-5L) Visual Analogue Scale (VAS) Score at Baseline, Week 12, 24 and 52
Description: EQ-5D-5L: Standardized, participant-rated questionnaire to assess health-related quality of life. EQ-5D-5L includes 2 components: EQ-5D-5L health state profile (descriptive system) and EQ-5D-5L Visual Analog Scale. EQ-5D-5L descriptive system provides a profile of participant's health state 5 dimensions:
  mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response options (no problems, slight problems, moderate problems, severe problems and extreme problems) that reflect increasing levels of difficulty. Responses to 5 dimension scores were combined and converted into single preference-weighted health utility index score 0 (worst health state) to 1 (better health state). EQ-VAS: Self-rated health status using a vertical VAS. EQ-VAS records participant's perceptions of their own current overall health in range from 0 (worst imaginable health) to 100 (best imaginable health).
Time Frame: Baseline, Week 12, 24 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Units on a scale
  Baseline: number analyzed (Participants) | 134 | 133
  Baseline | 42.4 (18.5) | 45.4 (20.4)
  Week 12: number analyzed (Participants) | 142 | 140
  Week 12 | 64.6 (19.6) | 63.2 (20.9)
  Week 24: number analyzed (Participants) | 139 | 132
  Week 24 | 66.2 (22.2) | 65.6 (24.3)
  Week 52: number analyzed (Participants) | 121 | 118
  Week 52 | 68.8 (21.7) | 69.0 (22.7)

23. Secondary Outcome: Mean Change From Baseline (Week 4) in Injection Site Pain as Assessed by Visual Analogue Scale (VAS) at Week 6 and 8
Description: The participant's reported perception of pain was measured on a VAS where the slash drawn by the participant represents pain of increasing intensity. VAS score ranges from 0-10 millimeter [mm], where; 0 mm=no pain and 10 mm=worst possible pain. The first 2 injections was administered by qualified personnel. The next three doses of IMP (3-5) will be self-administered by the participant and injection site pain was assessed. Pain was recorded immediately after, 15 minutes after, and 1 hour after the injections received by the participants.
Time Frame: Immediately, 15 minutes and 1 hour post-injection on Baseline (Week 4), Week 6 and 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | MSB11022 | EU-Humira
Number analyzed (Participants) | 143 | 145
Millimeter (mm)
  Change at Week 6: Immediately post-injection: number analyzed (Participants) | 140 | 143
  Change at Week 6: Immediately post-injection | -1.4 (5.12) | -1.3 (10.16)
  Change at Week 6: 15 min post-injection: number analyzed (Participants) | 140 | 143
  Change at Week 6: 15 min post-injection | -0.2 (2.67) | 0.4 (3.29)
  Change at Week 6: 1 hour post-injection: number analyzed (Participants) | 140 | 143
  Change at Week 6: 1 hour post-injection | 0.0 (0.66) | 0.0 (2.67)
  Change at Week 8: Immediately post-injection: number analyzed (Participants) | 140 | 139
  Change at Week 8: Immediately post-injection | -1.7 (6.48) | -2.3 (10.35)
  Change at Week 8: 15 min post-injection: number analyzed (Participants) | 140 | 139
  Change at Week 8: 15 min post-injection | -0.3 (2.25) | -0.7 (4.12)
  Change at Week 8: 1 hour post-injection: number analyzed (Participants) | 140 | 139
  Change at Week 8: 1 hour post-injection | -0.1 (0.57) | -0.7 (5.43)

ADVERSE EVENTS:
Time Frame: Up to Week 69
Arm/Group | MSB11022 | EU-Humira
All-Cause Mortality (participants affected / at risk) | 0/143 | 2/145
Serious Adverse Events (participants affected / at risk) | 8/143 | 15/145
Other Adverse Events (participants affected / at risk) | 15/143 | 34/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSB11022 (N=143) | EU-Humira (N=145)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Mycobacterium tuberculosis complex test positive (Investigations) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 1 | 0
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Death (General disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MSB11022 (N=143) | EU-Humira (N=145)
Injection site erythema (General disorders) | 4 | 12
Injection site pain (General disorders) | 2 | 10
Injection site pruritus (General disorders) | 1 | 8
Nasopharyngitis (Infections and infestations) | 6 | 13
Erythema (Skin and subcutaneous tissue disorders) | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT03052322/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT03052322/SAP_001.pdf